CLINICAL TRIAL: NCT06768697
Title: Safety and Immunogenicity Evaluation of the Recombinant Flagellin Protein Adjuvant in the SARS-CoV-2 Subunit Mucosal Vaccine
Brief Title: Safety and Immunogenicity Evaluation of the Recombinant Flagellin Protein Adjuvant
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shanghai Public Health Clinical Center (Other Government)
Responsible Party: Principal Investigator, wu qingguo, associate chief physician, Shanghai Public Health Clinical Center
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2024-S084-02
Record Dates: First submitted 2024-12-23; First posted 2025-01-10 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: COVID - 19
Keywords: adjuvant; novel adjuvant; flagellin; mucosal vaccine; SARS-CoV-2
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group A (Experimental): A total of 15 participants were enrolled, with 12 receiving the KFD1+3R-NC (0µg + 80µg) nasal spray and 3 receiving the PBS nasal spray as a placebo control.
  Interventions: Biological: KFD1(0µg )
- Group B (Experimental): A total of 15 participants were enrolled, with 12 receiving the KFD1+3R-NC (20µg + 80µg) nasal spray and 3 receiving the PBS nasal spray as a placebo control .
  Interventions: Biological: KFD1(20µg)
- Group C (Experimental): A total of 15 participants were enrolled, with 12 receiving the KFD1+3R-NC (40µg + 80µg) nasal spray and 3 receiving the PBS nasal spray as a placebo control.
  Interventions: Biological: KFD1(40µg)
- Group D (Experimental): A total of 15 participants were enrolled, with 12 receiving the KFD1+3R-NC (80µg + 80µg) nasal spray and 3 receiving the PBS nasal spray as a placebo control.
  Interventions: Biological: KFD1(80µg)

INTERVENTIONS:
Biological: KFD1(0µg ) — SARS-CoV-2 subunit mucosal vaccine adjuvanted with flagellin protein(0µg + 80µg)
  Arms: Group A
Biological: KFD1(20µg) — SARS-CoV-2 subunit mucosal vaccine adjuvanted with flagellin protein(20µg + 80µg)
  Arms: Group B
Biological: KFD1(40µg) — SARS-CoV-2 subunit mucosal vaccine adjuvanted with flagellin protein(40µg + 80µg)
  Arms: Group C
Biological: KFD1(80µg) — SARS-CoV-2 subunit mucosal vaccine adjuvanted with flagellin protein(80µg + 80µg)
  Arms: Group D

SUMMARY:
The goal of this clinical trial is to learn if the SARS-CoV-2 subunit mucosal vaccine with the recombinant flagellin protein adjuvant works to Prevent COVID-19 infection. It will also learn about the Safety and immunogenicity of the vaccine.

DETAILED DESCRIPTION:
This study explored the dosing of the 3R-NC containing BA.2.86 strain, EG.5 strain, and WIV 1 strain receptor binding domain（RBD） with the the recombinant flagellin protein adjuvant KFD1 （KFD1）in healthy subjects, further evaluating the safety, tolerability, and immunogenicity of the recombinant flagellin protein adjuvant KFD1 （KFD1） as a mucosal immune enhancer. KFD1 was divided into four dosage groups (0μg, 20μg, 40μg, 80μg), with each dosage group receiving two administrations. Safety assessments were conducted 7 days after each dosage group, and the next dosage group could only be administered after confirming safety. Samples including saliva, nasal wash, and blood were collected at different time points after the two vaccinations to evaluate safety and immunogenicity.

ELIGIBILITY:
Inclusion Criteria:

1. The subjects are healthy individuals aged between 18 and 65 years old (inclusive), with no gender preference, ensuring an appropriate gender ratio.
2. Have received 2-3 doses of COVID-19 inactivated vaccine, and the last dose was administered more than 6 months ago.
3. Have not been infected with COVID-19 within 3 months.
4. Capable of being used in conjunction with nasal sprays, and also suitable for nasal irrigation, saliva collection, and blood collection.
5. Male subjects and their partners, or female subjects, must agree to adopt one or more non-drug contraceptive measures (such as complete abstinence, condoms, intrauterine devices, partner sterilization, etc.) during the trial period and for six months after the trial ends, and they must not have plans for sperm donation or egg donation.
6. The subjects fully understand the purpose, nature, methods, and possible adverse reactions of the trial, voluntarily participate in the trial, and sign the informed consent form.
7. The subject is able to communicate effectively with the researcher and complete the study in accordance with the protocol.

Exclusion Criteria:

1. Active or suspected viral, bacterial, fungal, or parasitic infections, including herpes, shingles, or cold sores, within 14 days prior to screening.
2. History of recurrent infections of unknown causes; or use of systemic antibiotics within 90 days prior to drug administration.
3. Individuals with malignant tumors or a history of malignant tumors, except for non-melanoma skin cancer that has been cured for more than 3 years.
4. Nasal malformation, trauma, or other reasons that make it impossible to use nasal sprays.
5. Individuals with a history of allergy to biological agents or any drug components; individuals with a history of allergies, such as asthma, aspergillus infection, allergic rhinitis, etc., who have been determined by researchers to be unsuitable for enrollment.
6. Screen for outpatient or inpatient history of clinically significant chronic or acute disease symptoms within the previous 3 months, and ensure no surgical plans during the study period.
7. Previous tests have found HIV-Ab positive, HCV positive, and anti-syphilis helical-specific antibody positive (please consult the subject).
8. Individuals with abnormal vital signs (refer to normal range: systolic blood pressure 90~139mmHg, diastolic blood pressure 60~89mmHg, pulse rate 55-100 beats/min; body temperature (ear temperature) 35.4-37.7℃; respiratory rate 16-20 breaths/min) or abnormal electrocardiogram (QTcB≥450 ms, QTcB= QT/RR0.5) or clinically significant abnormalities in physical examination, laboratory tests (subject to the judgment of the clinical research doctor).
9. Screen for the use of other medications, including prescription or non-prescription drugs, and herbal remedies, within the previous 4 weeks.
10. Screen for individuals who have received vaccination within the previous 4 weeks or plan to receive vaccination during the study period.
11. Individuals with a history of significant allergic reactions (anaphylaxis or angioedema) to any products (such as food and drugs), and known to be allergic to the test drug, its excipients, or similar drugs.
12. Participate in any other drug clinical trials within 3 months before screening or within 5 half-lives of other clinical trial drugs (choose the longer time period).
13. Exclude individuals who have donated plasma or whole blood exceeding 200 mL within the previous 3 months, except during menstruation.
14. Individuals who abuse drugs or have used soft drugs (such as marijuana) within the past 3 months, or have consumed hard drugs (such as cocaine, phencyclidine, etc.) within the year prior to the trial; or individuals who test positive for drug abuse in urine screening (including methamphetamine, ketamine, MDMA, marijuana, morphine).
15. Individuals who are alcoholics or have regularly consumed alcohol within the 6 months prior to the trial, with an average weekly alcohol intake exceeding 14 units (1 unit of alcohol is equivalent to approximately 360 mL of beer, 45 mL of spirits with a 40% alcohol content, or 150 mL of wine), or those who cannot abstain from alcohol during the trial period (interview).
16. Subjects who have smoked an average of more than 5 cigarettes per day or used other nicotine-containing products (such as nicotine patches, nicotine gum, e-cigarettes, etc.) more than 5 times per day on average within the previous 3 months, or who cannot stop using any tobacco-related products during the trial period.
17. Those who have previously or currently suffered from any clinically severe diseases of the circulatory system, endocrine system, nervous system, digestive system, respiratory system, urogenital system, hematology, immunology, psychiatry, or metabolic abnormalities, or any other diseases that may interfere with the results of the trial.
18. Use other medications, including prescription or non-prescription drugs, and Chinese herbal medicine, from the screening date to D1.
19. Women who are pregnant, breastfeeding, or may become pregnant.
20. Clinical diagnosis of any autoimmune disease or rheumatic disease.
21. The patient's blood COVID-19 specific IgG antibody is greater than 1×10e4.
22. Any situation that other researchers consider unsuitable for participation in the study.

    -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-12-30 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Safety Tolerance Evaluation Indicators | Screening period, Day1, Day2, Day22、Day23、Day43±2
  Evaluate the adverse reactions of patients after vaccination according to the CTCAE standards, which include local reactions and systemic reactions, graded from level 1 to level 5.

SECONDARY OUTCOMES:
IgA and IgG titers in saliva and nasal wash fluid | saliva：Day1、Day22、Day43±2、Day112±5、Day202±5；nasal wash fluid：Day1、Day22、Day43±2、Day112±5、Day202±5
  Using the ELISA method, we detected RBD-specific IgA, IgG, as well as total IgA and IgG titers in saliva and nasal wash samples, and calculated the relative concentrations of RBD-specific IgA and IgG in total IgA and IgG.
plasma SARS-CoV-2 RBD-specific IgG and IgA titers | Screening period, Day1、Day22、Day43±2、Day112±5、Day202±5
  Determination of Plasma SARS-CoV-2 RBD-Specific IgG, IgA Titers
plasma neutralizing antibody titers | Day1、Day22、Day43±2、Day112±5、Day202±5
  Using the ELISA method, we detected plasma neutralizing antibody titers
Titers of flagellin-specific IgG and IgA in plasma | Day1、Day22、Day43±2、Day112±5、Day202±5
  Determination of flagellin-specific IgG and IgA in plasma

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Public Health Clinical Center,Fudan University, Shanghai, Jinshan District, China

IPD SHARING:
Plan to Share IPD: Yes
If you need to view it, you can apply to the applicant for access.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: From December 2025 to December 2026
Access Criteria: Research information can be obtained after obtaining authorization from the researcher